CLINICAL TRIAL: NCT01661621
Title: Antimuscarinics as the First-line Treatment for Male With International Prostate Symptom Score (IPSS) Voiding-to-storage Subscore Rati (IPSS-V/S)≤1-- A Prospective Randomized Study Comparing With α-blockers
Brief Title: Antimuscarinics as the First-line Treatment for Male With IPSS-V/S≤1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hann-Chorng Kuo, Department of Urology, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCGHUROL002
Record Dates: First submitted 2012-08-02; First posted 2012-08-09 (Estimated); Results first posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Bladder Outlet Obstruction
Keywords: Lower urinary tract symptoms (LUTS); International Prostate Symptom Score (IPSS); Antimuscarinics; α-blockers
MeSH Terms: conditions — Urinary Bladder Neck Obstruction; Lower Urinary Tract Symptoms | interventions — Tolterodine Tartrate; Doxazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Antimuscarinics (Detrusitol 4 mg QD)
  Interventions: Drug: Detrusitol 4 mg QD
- Group 2 (Experimental): α-blockers (Doxazosin 4 mg QD)
  Interventions: Drug: Doxazosin 4 mg QD

INTERVENTIONS:
Drug: Detrusitol 4 mg QD — Group 1
  Arms: Group 1
Drug: Doxazosin 4 mg QD — Group 2
  Arms: Group 2

SUMMARY:
This study is a prospective randomized, open label, controlled, double arm, post-marketing study to compare the treatment efficacy of first-line antimuscarinics and α-blockers monotherapy for men with moderate to severe lower urinary tract symptoms (LUTS) (International Prostate Symptom Score (IPSS-T) ≥8) and IPSS voiding-to-storage subscore ratio (IPSS-V/S) ≤1.

DETAILED DESCRIPTION:
1. STUDY PROCEDURE

1.1.General Study Design This study is a prospective randomized, open label, controlled, double arm, post-marketing study to compare the treatment efficacy of first-line antimuscarinics and α-blockers monotherapy for men with moderate to severe LUTS (IPSS-T ≥8) and IPSS-V/S ≤1.

1.2. Study Visits and Evaluations

1.2.1 Screening Visit (Baseline, 1 day to 1 week of the first treatment day).

1.2.1.1 Explain the nature of the study and have patients to read and sign an Informed Consent Form.

1.2.1.2 Screen patients for inclusion/exclusion criteria. 1.2.1.3 Medical History of lower urinary tract symptoms and previous treatment modalities.

1.2.1.4 Vital signs monitoring, general physical examinations of all systems (including digital rectal examination), serum prostatic specific antigen (PSA), and urinalysis.

1.2.1.5 Record Patient Perception of Bladder Condition (PPBC), IPSS (IPSS-T, IPSS voiding (IPSS-V), and IPSS storage (IPSS-S)), Overactive Bladder Symptom Score (OAB-SS), and quality of Life index (QoL-I)scores.

1.2.1.6 Obtain maximum flow rate (Qmax), voided volume, postvoid residual volume (PVR), total prostate volume (TPV), and transitional zone index (TZI).

1.2.1.7 Randomized assigned patients into 2 groups; men in one group received Doxazosin 4 mg QD, and those in the other group received Detrusitol 4 mg QD.

1.2.2 First Evaluation Visit (2 weeks after the initial treatment) 1.2.2.1 Vital signs monitoring and record adverse events. 1.2.2.2 Record PPBC, IPSS (IPSS-T, IPSS-V, IPSS-S), OAB-SS and QoL. 1.2.2.3 Check urinalysis for urinary tract infection if patient has symptoms suggestive of urinary tract infection.

1.2.2.4 Check Qmax, voided volume, and PVR.

1.2.3 Second Evaluation Visit (4 weeks after the treatment). 1.2.3.1 Vital signs monitoring and record adverse events. 1.2.3.3 Check urinalysis for urinary tract infection if patient has symptoms suggestive of urinary tract infection.

1.2.3.4 Check Qmax, voided volume, and PVR.

1.2.4 Third Evaluation Visit (3 months after the treatment). 1.2.4.1 Vital signs monitoring and record adverse events. 1.2.4.2 Record PPBC, IPSS (IPSS-T, IPSS-V, IPSS-S), OAB-SS and QoL. 1.2.4.3 Check urinalysis for urinary tract infection if patient has symptoms suggestive of urinary tract infection.

1.2.4.4 Check Qmax, voided volume, and PVR.

1.3. Withdrawal Criteria

Patients with any of the following conditions may be withdrawn from the trial:

1.3.1. Patients decide to withdraw their consent. 1.3.2. Patients indicate the status of lack of efficacy which is of clinical significance judged by the investigators that may lead to permanent damage to the patients.

1.3.3. Investigators consider that there is of safety concerns for the patients to remain in the trial (such as development severe medical disease).

1.3.4. Lost of follow-up or death. 1.3.5. PVR≥300 mL

1.4. Concomitant Treatments Investigator will try to minimize the concomitant medications for the patients during the trial duration. However, patients are allowed to continue taking stable medication in stable dose for diseases other than genitourinary system.

1.5. Prohibited medication

Patients are not allowed to take any of the following medications during the study:

1. Anticholinergics other than test drug
2. Alpha-adrenergic receptor blockers
3. Tricyclic anti-depressants
4. Calcium channel blockers
5. Skeletal muscle relaxant
6. Cyclooxygenase-2 (COX-2) inhibitors

ELIGIBILITY:
Inclusion Criteria:

* Men aged ≥40 years with lower urinary tract symptoms (IPSS ≥8)
* Patient or his/her legally acceptable representative has signed the written informed consent form

Exclusion Criteria:

* Patients with severe cardiopulmonary disease and such as congestive heart failure, arrhythmia, poorly controlled hypertension, not able to receive regular follow-up
* Patients with urinary retention, urodynamically proven detrusor underactivity or PVR ≥250 mL
* Patients with known active urinary tract infection, urinary stone or malignancy
* Patients with history of urethral injury or transurethral surgery for prostate or bladder
* Patients have laboratory abnormalities at screening including:

  1. Aspartate aminotransferase (AST) >3 x upper limit of normal range
  2. Alanine aminotransferase (ALT) >3 x upper limit of normal range
  3. Patients have abnormal serum creatinine level >2 x upper limit of normal range
* Patients with any other serious disease or condition considered by the investigator not suitable for entry into the trial
* Patients participated investigational drug trial within 1 month before entering this study
* Patients with major psychiatric illness or drug abuse
* Patients taken medication such as alpha-blocker, antimuscarinic or 5 alpha-reductase (5AR) inhibitor within 6 months

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hann-Chorng Kuo, M.D., Principal Investigator — Department of Urology, Buddhist Tzu Chi General Hospital and Tzu Chi University
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

REFERENCES:
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Background] Chapple CR, Roehrborn CG. A shifted paradigm for the further understanding, evaluation, and treatment of lower urinary tract symptoms in men: focus on the bladder. Eur Urol. 2006 Apr;49(4):651-8. doi: 10.1016/j.eururo.2006.02.018. Epub 2006 Feb 17. PMID 16530611
- [Background] Athanasopoulos A, Gyftopoulos K, Giannitsas K, Fisfis J, Perimenis P, Barbalias G. Combination treatment with an alpha-blocker plus an anticholinergic for bladder outlet obstruction: a prospective, randomized, controlled study. J Urol. 2003 Jun;169(6):2253-6. doi: 10.1097/01.ju.0000067541.73285.eb. PMID 12771763
- [Background] Lee JY, Kim HW, Lee SJ, Koh JS, Suh HJ, Chancellor MB. Comparison of doxazosin with or without tolterodine in men with symptomatic bladder outlet obstruction and an overactive bladder. BJU Int. 2004 Oct;94(6):817-20. doi: 10.1111/j.1464-410X.2004.05039.x. PMID 15476515
- [Background] Kaplan SA, Roehrborn CG, Rovner ES, Carlsson M, Bavendam T, Guan Z. Tolterodine and tamsulosin for treatment of men with lower urinary tract symptoms and overactive bladder: a randomized controlled trial. JAMA. 2006 Nov 15;296(19):2319-28. doi: 10.1001/jama.296.19.2319. PMID 17105794
- [Background] Kaplan SA, McCammon K, Fincher R, Fakhoury A, He W. Safety and tolerability of solifenacin add-on therapy to alpha-blocker treated men with residual urgency and frequency. J Urol. 2009 Dec;182(6):2825-30. doi: 10.1016/j.juro.2009.08.023. Epub 2009 Oct 17. PMID 19837435
- [Background] Chung DE, Te AE, Staskin DR, Kaplan SA. Efficacy and safety of tolterodine extended release and dutasteride in male overactive bladder patients with prostates >30 grams. Urology. 2010 May;75(5):1144-8. doi: 10.1016/j.urology.2009.12.010. Epub 2010 Mar 5. PMID 20206978
- [Background] Chung SD, Chang HC, Chiu B, Liao CH, Kuo HC. The efficacy of additive tolterodine extended release for 1-year in older men with storage symptoms and clinical benign proastatic hyperplasia. Neurourol Urodyn. 2011 Apr;30(4):568-71. doi: 10.1002/nau.20923. Epub 2011 Feb 22. PMID 21344494
- [Background] Blake-James BT, Rashidian A, Ikeda Y, Emberton M. The role of anticholinergics in men with lower urinary tract symptoms suggestive of benign prostatic hyperplasia: a systematic review and meta-analysis. BJU Int. 2007 Jan;99(1):85-96. doi: 10.1111/j.1464-410X.2006.06574.x. Epub 2006 Oct 9. PMID 17026588
- [Background] Martin-Merino E, Garcia-Rodriguez LA, Masso-Gonzalez EL, Roehrborn CG. Do oral antimuscarinic drugs carry an increased risk of acute urinary retention? J Urol. 2009 Oct;182(4):1442-8. doi: 10.1016/j.juro.2009.06.051. Epub 2009 Aug 15. PMID 19683302
- [Background] McVary KT, Roehrborn CG, Avins AL, Barry MJ, Bruskewitz RC, Donnell RF, Foster HE Jr, Gonzalez CM, Kaplan SA, Penson DF, Ulchaker JC, Wei JT. Update on AUA guideline on the management of benign prostatic hyperplasia. J Urol. 2011 May;185(5):1793-803. doi: 10.1016/j.juro.2011.01.074. Epub 2011 Mar 21. PMID 21420124
- [Background] Djavan B, Margreiter M, Dianat SS. An algorithm for medical management in male lower urinary tract symptoms. Curr Opin Urol. 2011 Jan;21(1):5-12. doi: 10.1097/MOU.0b013e32834100ef. PMID 21045704
- [Background] Kaplan SA, Roehrborn CG, Abrams P, Chapple CR, Bavendam T, Guan Z. Antimuscarinics for treatment of storage lower urinary tract symptoms in men: a systematic review. Int J Clin Pract. 2011 Apr;65(4):487-507. doi: 10.1111/j.1742-1241.2010.02611.x. Epub 2011 Jan 7. PMID 21210910
- [Background] Athanasopoulos A, Chapple C, Fowler C, Gratzke C, Kaplan S, Stief C, Tubaro A. The role of antimuscarinics in the management of men with symptoms of overactive bladder associated with concomitant bladder outlet obstruction: an update. Eur Urol. 2011 Jul;60(1):94-105. doi: 10.1016/j.eururo.2011.03.054. Epub 2011 Apr 9. PMID 21497434
- [Background] Chapple C. Antimuscarinics in men with lower urinary tract symptoms suggestive of bladder outlet obstruction due to benign prostatic hyperplasia. Curr Opin Urol. 2010 Jan;20(1):43-8. doi: 10.1097/MOU.0b013e3283330862. PMID 19875964
- [Background] Liao CH, Chung SD, Kuo HC. Diagnostic value of International Prostate Symptom Score voiding-to-storage subscore ratio in male lower urinary tract symptoms. Int J Clin Pract. 2011 May;65(5):552-8. doi: 10.1111/j.1742-1241.2011.02638.x. PMID 21489080

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 116 | 279
Completed | 116 | 279
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 116 | 279 | 395
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (11.3) | 65.6 (10.5) | 66.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 116 | 279 | 395
Region of Enrollment [Number; unit: participants]
  Taiwan | 116 | 279 | 395

OUTCOME MEASURES:

1. Primary Outcome: The Global Response Assessment (GRA) After the Treatment Day
Description: Efficacy Using global response assessment (GRA) to compare the efficacy in Group 1 and Group 2 from baseline to 1month.
  The global response assessment on a 6-point scale ranging from 1 "No problems at all" to 6 "Many severe problems".
  Changes of the global response assessment (GRA) improved or reduction by 1 points.
  Change = Baseline minus Month 1 value
  Safety:
  Systemic adverse events such as difficult urination, dry mouth, dry eye, blurred vision, constipation, dizziness or general weakness
Time Frame: 1 month after initial treatment
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 116 | 279
participants
  GRA≥1 | 89 | 218
  GRA<1 | 27 | 61

2. Secondary Outcome: The International Prostate Symptom Score (IPSS) Questionnaires After the Treatment Day
Description: Efficacy:
  Using the total International Prostate Symptom Score (IPSS) to compare the efficacy in Group 1 and Group 2 from baseline to 1 month.
  The International Prostate Symptom Score (IPSS) is an 7 symptom questions including 4 voiding questions (IPSS-voiding), 3 storage questions (IPSS-Storage) The symptom score have 6-point scale ranging from 0 "Not at all" to 5 "Almost always".
  Total IPSS score = IPSS-voiding + IPSS-Storage Rang = 0 to 35 (asymptomatic to very symptomatic). Mild = 0 to 7; Moderate = 8 to 19; Severe = 20 to 35
  Safety:
  Systemic adverse events such as difficult urination, dry mouth, blurred vision, constipation, dry eye, dizziness, or general weakness
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 116 | 279
units on a scale
  Baseline | 14.8 (5.40) | 18.0 (6.47)
  1 month | 11.2 (6.81) | 10.8 (6.36)

3. Secondary Outcome: The Maximum Flow Rate (Qmax) After the Treatment Day
Description: Efficacy:
  Net change used the the maximum flow rate (Qmax) in Group 1 and Group 2 from baseline to 1 month.
  Safety:
  Systemic adverse events such as difficult urination, dry mouth, blurred vision, constipation, dry eye, dizziness, or general weakness
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: mL/s
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 116 | 279
mL/s
  Baseline | 13.1 (8.10) | 11.4 (5.95)
  1 month | 13.6 (7.90) | 13.6 (6.63)

4. Secondary Outcome: The Voided Volume After the Treatment Day
Description: Efficacy:
  Net change used the the voided volume in Group 1 and Group 2 from baseline to 1 month.
  Safety:
  Systemic adverse events such as difficult urination, dry mouth, blurred vision, constipation, dry eye, dizziness, or general weakness
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 116 | 279
mL
  Baseline | 212.5 (168.8) | 244.0 (148.3)
  1 month | 231.6 (163.6) | 268.3 (150.7)

5. Secondary Outcome: The Postvoid Residual Volume (PVR) After the Treatment Day
Description: Efficacy:
  Net change used the the postvoid residual volume (PVR) in Group 1 and Group 2 from baseline to 1 month.
  Safety:
  Systemic adverse events such as difficult urination, dry mouth, blurred vision, constipation, dry eye, dizziness, or general weakness
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 116 | 279
mL
  Baseline | 50.1 (62.6) | 53.9 (58.7)
  1 month | 60.4 (60.4) | 42.9 (49.3)

6. Secondary Outcome: The IPSS Subscore (IPSS Voiding) Questionnaires After the Treatment Day
Description: Efficacy:
  Using the the IPSS subscore (IPSS Voiding) questionnaires to compare the efficacy in Group 1 and Group 2 from baseline to 1 month.
  The IPSS subscore (IPSS Voiding) questionnaires is a 4 symptom questions. The symptom score have 6-point scale ranging from 0 "Not at all" to 5 "Almost always". Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom.
  The total IPSS Voiding score can therefore range from 0 to 20 (asymptomatic to very symptomatic).
  Safety:
  Systemic adverse events such as difficult urination, dry mouth, blurred vision, constipation, dry eye, dizziness, or general weakness
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 116 | 279
units on a scale
  Baseline | 5.31 (3.51) | 12.3 (4.37)
  1 month | 4.84 (4.75) | 6.49 (4.97)

7. Secondary Outcome: The IPSS Subscore (IPSS Storage) Questionnaires After the Treatment Day
Description: Efficacy:
  Using the the IPSS subscore (IPSS Storage) to compare the efficacy in Group 1 and Group 2 from baseline to 1 month.
  The IPSS subscore (IPSS Storage) is a 3 symptom questions. The symptom score have 6-point scale ranging from 0 "Not at all" to 5 "Almost always". Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom.
  The total IPSS Storage score can therefore range from 0 to 15 (asymptomatic to very symptomatic).
  Safety:
  Systemic adverse events such as difficult urination, dry mouth, blurred vision, constipation, dry eye, dizziness, or general weakness
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 116 | 279
units on a scale
  Baseline | 9.51 (3.05) | 5.70 (3.09)
  1 month | 6.40 (3.47) | 4.31 (2.80)

8. Secondary Outcome: The International Prostate Symptom Score (IPSS) Quality of Life (QoL) Score After the Treatment Day
Description: Efficacy:
  Using the the the International Prostate Symptom Score (IPSS) quality of life (QoL) score to compare the efficacy in Group 1 and Group 2 from baseline to 1month.
  The IPSS quality of life question score on a 7-point scale ranging from 0 "Delighted" to 6 "Terrible".
  IPSS-QoL ranges 0 to 6 (Delighted to Terrible)
  Safety:
  Systemic adverse events such as difficult urination, dry mouth, blurred vision, constipation, dry eye, dizziness, or general weakness
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 116 | 279
units on a scale
  Baseline | 3.91 (1.01) | 3.88 (0.82)
  1 month | 2.82 (1.18) | 2.82 (0.96)

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/279
Other Adverse Events (participants affected / at risk) | 18/116 | 33/279
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=116) | Group 2 (N=279)
Dizziness (General disorders) | 12 | 0
General weakness (General disorders) | 3 | 0
Palpitation (General disorders) | 3 | 0
Dry mouth (General disorders) | 0 | 13
Blurred vision (General disorders) | 0 | 10
Dry eye (General disorders) | 0 | 7
Constipation (General disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes